CLINICAL TRIAL: NCT05463354
Title: Safety and Immunogenicity of Recombinant COVID-19 Vaccine (Sf9 Cell) as a Booster Following Primary Vaccination of Either Inactivated or mRNA or Viral Vector COVID-19 Vaccines
Brief Title: Safety and Immunogenicity of Recombinant COVID-19 Vaccine (Sf9 Cell) as a Booster
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: WestVac Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: WSTVC001
Record Dates: First submitted 2022-07-18; First posted 2022-07-19 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Inactivated COVID-19 vaccines cohort group 1 (Experimental): Participants who received 2 doses of Inactivated COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment. N=75 Intervention: Recombinant COVID-19 Vaccine (Sf9 Cell)
  Interventions: Biological: Recombinant COVID-19 Vaccine (Sf9 Cell)
- Inactivated COVID-19 vaccines cohort group 2 (Active Comparator): Participants who received 2 doses of Inactivated COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment. N=75 Intervention: COVID-19 Vaccine (Vero Cell), Inactivated
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- mRNA COVID-19 vaccines cohort group 1 (Experimental): Participants who received 2 doses of mRNA COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment. N=75 Intervention: Recombinant COVID-19 Vaccine (Sf9 Cell)
  Interventions: Biological: Recombinant COVID-19 Vaccine (Sf9 Cell)
- mRNA COVID-19 vaccines cohort group 2 (Active Comparator): Participants who received 2 doses of mRNA COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment. N=75 Intervention: COVID-19 Vaccine (Vero Cell), Inactivated
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- Viral Vector COVID-19 vaccines cohort group 1 (Experimental): Participants who received 2 doses of Viral Vector COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment. N=75 Intervention: Recombinant COVID-19 Vaccine (Sf9 Cell)
  Interventions: Biological: Recombinant COVID-19 Vaccine (Sf9 Cell)
- Viral Vector COVID-19 vaccines cohort group 2 (Active Comparator): Participants who received 2 doses of Viral Vector COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment. N=75 Intervention: COVID-19 Vaccine (Vero Cell), Inactivated
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated

INTERVENTIONS:
Biological: Recombinant COVID-19 Vaccine (Sf9 Cell) — 1dose, Intramuscular Injection
  Arms: Inactivated COVID-19 vaccines cohort group 1; Viral Vector COVID-19 vaccines cohort group 1; mRNA COVID-19 vaccines cohort group 1
Biological: COVID-19 Vaccine (Vero Cell), Inactivated — 1dose, Intramuscular Injection
  Arms: Inactivated COVID-19 vaccines cohort group 2; Viral Vector COVID-19 vaccines cohort group 2; mRNA COVID-19 vaccines cohort group 2

SUMMARY:
A phase Ⅱ, observer-blind, randomized, controlled, investigator-initiated clinical trial to evaluate the safety and immunogenicity of a booster vaccination with Recombinant COVID-19 vaccine (Sf9 Cell) in a population aged 18 years and above who have completed homologous primary vaccination with either Inactivated or mRNA or Viral Vector COVID-19 vaccines at least 6 months prior to enrolment.

DETAILED DESCRIPTION:
A phase Ⅱ, observer-blind, randomized, controlled, investigator-initiated clinical trial to evaluate the safety and immunogenicity of a booster vaccination with Recombinant COVID-19 vaccine (Sf9 Cell) in a population aged 18 years and above who have completed homologous primary vaccination with either Inactivated or mRNA or Viral Vector COVID-19 vaccines at least 6 months prior to enrolment. The study uses a non-inferiority design to compare between schedules with Recombinant COVID-19 Vaccine (Sf9 Cell) versus COVID-19 Vaccine (Vero Cell), Inactivated as the booster dose. Participants, laboratory and analysing statisticians will remain blind to treatment allocation.

A total of 450 participants will be enrolled (participants aged ≥ 60 years account for approximately 10%), consisting of 3 cohorts:

150 participants who received 2 doses of Inactivated COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment.

150 participants who received 2 doses of mRNA COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment.

150 participants who received 2 doses of Viral Vector COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment.

Each of 3 cohorts of 150 participants will be randomized 1:1 to receive a single dose of Recombinant COVID-19 vaccine (Sf9 Cell) (test group) or the COVID-19 Vaccine (Vero Cell), Inactivated (control group).

ELIGIBILITY:
Inclusion Criteria:

* 1. Participant is willing and able to give written informed consent for participation in the trial.
* 2. Male or Female, aged 18 years or above and in good health as determined by a trial clinician.
* 3. Female participants of childbearing potential must be willing to ensure that they or their partner use effective contraception from 1 month prior to first immunisation continuously until 3 months after boost immunisation. See Section "Contraception and Pregnancy" for definition of child-bearing potential and definition of effective contraception.
* 4. In the Investigator's opinion, is able and willing to comply with all trial requirements.
* 5. Willing to allow investigators to discuss the volunteer's medical history with their General Practitioner and access all medical records when relevant to study procedures.
* 6. Agreement to refrain from blood donation during the study.
* 7. Participants who have completed homologous primary vaccination with either Inactivated or mRNA or Viral Vector COVID-19 vaccines (full approval, CMA or EUA) and is at least 6 months post second vaccination.

Exclusion Criteria:

* 1. Receipt of any vaccine (licensed or investigational) other than the study intervention within 30 days before and after each study vaccination (one week for licensed seasonal influenza vaccine or pneumococcal vaccine)
* 2. Prior or planned receipt of any other investigational or licensed vaccine or product likely to impact on interpretation of the trial data (e.g. adenovirus vectored vaccines, any coronavirus vaccines)
* 3. Positive SARS-CoV-2 RT-PCR at screening.
* 4. Participants who are pregnant at enrolment or planning to become pregnant during the first 3 months following vaccination.
* 5. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccines.
* 6. Any confirmed or suspected immunosuppressive or immunodeficient state; asplenia; recurrent severe infections and use of immunosuppressant medication within the past 6 months, except topical steroids or short-term oral steroids (course lasting ≤14 days).
* 7. History of allergic disease or reactions likely to be exacerbated by any component of study vaccines.
* 8. Any history of anaphylaxis.
* 9. Current diagnosis of or treatment for cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions (ADRs) | Day 0-28 post-boost dose.
Geometric mean titer (GMT) of specific neutralizing antibody (Virus or Pseudovirus Neutralization Assay) against SARS-CoV-2 | Day 14 post-boost dose.
Seroconversion rate (≥ 4 folds increase from baseline) of serum anti-SARS-CoV-2 neutralizing antibody titers | Day 14 post-boost dose.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Day 0-7 post-boost dose
Incidence of AEs | Day 0-28 post-boost dose
Incidence of serious adverse events (SAEs) | Day 0 through 6 months post-boost dose
The percentage of participants with abnormal hematology, chemistry and urinalysis laboratory values | Day 3 post-boost dose
The percentage of participants with grading shifts in hematology, chemistry and urinalysis laboratory assessments between baseline and 3 days after the booster dose. | Day 3 post-boost dose
GMT of specific neutralizing antibody (Virus or Pseudovirus Neutralization Assay) against SARS-CoV-2 | Day 28, month 3 and month 6 post-boost dose
Geometric mean increase (GMI) of specific neutralizing antibody (Virus or Pseudovirus Neutralization Assay) against SARS-CoV-2 | Day 14, day 28, month 3 and month 6 post-boost dose
GMT and GMI of IgG antibodies against SARS-CoV-2 S protein RBD | Day 14, day 28, month 3 and month 6 post-boost dose

CONTACTS AND LOCATIONS:
Locations (1):
- Iloilo Doctors Hospital, Iloilo City, Philippines